CLINICAL TRIAL: NCT01809106
Title: RCT Comparing the Analgesic Efficacy of 4 Therapeutic Strategies Based on 4 Different Major Opioids (Fentanyl, Oxycodone, Buprenorphine vs Morphine) in Cancer Patients With Moderate/Severe Pain, at the Moment of Starting 3rd Step of WHO Analgesic Ladder.
Acronym: CERP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Studio CERP
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-10

CONDITIONS: Cancer; Cancer Pain
Keywords: cancer pain; major opioid; analgesics
MeSH Terms: conditions — Neoplasms; Cancer Pain | interventions — Morphine; Fentanyl; Buprenorphine; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Morphine (Active Comparator)
  Interventions: Drug: Morphine
- Oxycodone (Experimental)
  Interventions: Drug: Oxycodone
- Buprenorphine (Experimental)
  Interventions: Drug: Buprenorphine
- Fentanyl (Experimental)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Morphine — 60 mg /24 ore
  Arms: Morphine
Drug: Fentanyl — 25 microg/h
  Arms: Fentanyl
Drug: Buprenorphine — 35 microg/h
  Arms: Buprenorphine
Drug: Oxycodone — 40 mg /24 ore
  Arms: Oxycodone

SUMMARY:
Pain, in neoplastic disease, is a symptom with severe negative impact on the quality of life of patients and a high incidence, with values around 70-90% in advanced and metastatic stages. Than 20 years the main reference for the pharmacological treatment of cancer pain are the guidelines produced by the World Health Organization (WHO). This document shows that the use of opioid drugs is the mainstay of treatment, with particular reference to opioids "major" (3 rd step of the analgesic ladder). The 4 opioids more most commonly prescribed in Italy (oral morphine and oxycodone, fentanyl and buprenorphine transdermal), based on the data currently available, have an analgesic effect would partly overlap but with different percentages of non-responders (NR), a different need to increase the dose over time to maintain adequate analgesia, a different action to the switch to another molecule for ineffectiveness analgesic. The observations described suggest that opioids, although they belong to the same family drug may not be fully comparable with regard to the clinical effects products. Important differences are known on the pharmacokinetic and pharmacodynamic and, more recently, also in terms of pharmacogenomics. This is a comparative study of analgesic strategies based on the use of the 4 mentioned opioids, going to look for possible differences in terms of analgesic efficacy, changes in dose over time, use of switch or permanent abandonment of treatment, parallel to the contour of the side effects. The associated sub-project will link the structure gene of patients and clinical results have emerged.

ELIGIBILITY:
Inclusion Criteria:

* patients with diagnostic (histological or cytological) evidence of locally advanced or metastatic solid tumour;
* with average pain intensity ≥ 4, measured with NRS and related to the last 24 hours, due to the cancer, requiring for the first time an analgesic treatment with 3rd step/WHO opioids
* with life expectancy > one month
* "strong" opioid naïve;
* eligible to take any of the medications under evaluation, by TDS or by mouth;
* with age ≥ 18 years;

Exclusion Criteria:

* Patients recruited in other researches that conflict or may confound the conduction and results of the present study;
* Lack of informed consent;
* with presence of other diseases, including psychiatric/mental illness, severe senile or other form of dementia, that can interfere with participation and compliance with the study protocol or can contraindicate the use of the investigational drugs;
* with presence of co-morbidities, which could create potentially dangerous drug interactions with opioids (eg, use of macrolide antibiotics or antifungal,….);
* any kind of contraindications to the use of opioid drugs;
* Patients with a known story, past or current, of drugs abuse or addiction;
* Use of drugs which presents a combination of opioids and other molecule (as NSAIDs, paracetamol, naloxone, ..);
* Patients who cannot guarantee regular follow-up visits for logistic or geographic reasons;
* Need of starting 3rd step treatment in an "emergency clinical situation" that do not allow the correct procedures of randomization;
* diagnosis of primary brain tumor or leukaemia;
* diagnosis of chronic renal failure;
* patients with antalgic radiotherapy or radio-metabolic therapy in progress or completed less than 14 days before study;
* patients starting a first line chemotherapy simultaneously to the beginning of the study;
* other types of analgesic treatments, including local-regional anesthetic techniques or neurosurgical /ablative methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2011-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Corli, MD, Principal Investigator — Mario Negri Institute of Pharmacological Research - IRCCS
Locations (9):
- Italy (9):
  - Ospedale S. Marta, Catania, Italy
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan, Italy
  - Istituto Scientifico San Raffaele, Milan, Italy
  - Azienda Ospedaliera Valtellina-Valchiavenna, Morbegno, Italy
  - Multimedica, Sesto San Giovanni, Italy
  - Ospedale Gradenigo, Torino, Italy
  - Ospedale Civile di Piacenza, Piacenza, Piacenza
  - Arcispedale S. Maria Nuova Azienda Ospedaliera, Reggio Emilia, RE
  - Ospedale San Giovanni Battista di Torino, Torino, Torino

REFERENCES:
- [Background] Apolone G, Bertetto O, Caraceni A, Corli O, De Conno F, Labianca R, Maltoni M, Nicora M, Torri V, Zucco F; Cancer Pain Outcome Research Study Group. Pain in cancer. An outcome research project to evaluate the epidemiology, the quality and the effects of pain treatment in cancer patients. Health Qual Life Outcomes. 2006 Feb 2;4:7. doi: 10.1186/1477-7525-4-7. PMID 16457716
- [Background] Apolone G, Corli O, Caraceni A, Negri E, Deandrea S, Montanari M, Greco MT; Cancer Pain Outcome Research Study Group (CPOR SG) Investigators. Pattern and quality of care of cancer pain management. Results from the Cancer Pain Outcome Research Study Group. Br J Cancer. 2009 May 19;100(10):1566-74. doi: 10.1038/sj.bjc.6605053. Epub 2009 Apr 28. PMID 19401688
- [Background] Greco MT, Corli O, Montanari M, Deandrea S, Zagonel V, Apolone G; Writing Protocol Committee; Cancer Pain Outcome Research Study Group (CPOR SG) Investigators. Epidemiology and pattern of care of breakthrough cancer pain in a longitudinal sample of cancer patients: results from the Cancer Pain Outcome Research Study Group. Clin J Pain. 2011 Jan;27(1):9-18. doi: 10.1097/AJP.0b013e3181edc250. PMID 20842024
- [Background] Apolone G, Deandrea S, Montanari M, Corli O, Greco MT, Cavuto S. Evaluation of the comparative analgesic effectiveness of transdermal and oral opioids in cancer patients: a propensity score analysis. Eur J Pain. 2012 Feb;16(2):229-38. doi: 10.1002/j.1532-2149.2011.00020.x. Epub 2011 Dec 19. PMID 22323375
- [Background] Corli O, Montanari M, Deandrea S, Greco MT, Villani W, Apolone G. An exploratory analysis on the effectiveness of four strong opioids in patients with cancer pain. Pain Med. 2012 Jul;13(7):897-907. doi: 10.1111/j.1526-4637.2012.01408.x. Epub 2012 Jun 8. PMID 22680789
- [Derived] Corli O, Roberto A, Bennett MI, Galli F, Corsi N, Rulli E, Antonione R. Nonresponsiveness and Susceptibility of Opioid Side Effects Related to Cancer Patients' Clinical Characteristics: A Post-Hoc Analysis. Pain Pract. 2018 Jul;18(6):748-757. doi: 10.1111/papr.12669. Epub 2018 Jan 17. PMID 29220110
- [Derived] Corli O, Floriani I, Roberto A, Montanari M, Galli F, Greco MT, Caraceni A, Kaasa S, Dragani TA, Azzarello G, Luzzani M, Cavanna L, Bandieri E, Gamucci T, Lipari G, Di Gregorio R, Valenti D, Reale C, Pavesi L, Iorno V, Crispino C, Pacchioni M, Apolone G; CERP STUDY OF PAIN GROUP (List of collaborators). Are strong opioids equally effective and safe in the treatment of chronic cancer pain? A multicenter randomized phase IV 'real life' trial on the variability of response to opioids. Ann Oncol. 2016 Jun;27(6):1107-1115. doi: 10.1093/annonc/mdw097. Epub 2016 Mar 2. PMID 26940689
- See also: Info of the study — http://crc.marionegri.it/cancerpain/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of First Enrollment: May 2014 Date of last enrollment: July 2014
Period: Overall Study
Arm/Group | Morphine | Oxycodone | Buprenorphine | Fentanyl
Started | 130 | 130 | 130 | 128
Completed | 122 | 125 | 127 | 124
Not Completed | 8 | 5 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morphine | Oxycodone | Buprenorphine | Fentanyl | Total
Number analyzed (Participants) | 122 | 125 | 127 | 124 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (11.7) | 66.9 (11.1) | 65.2 (13.5) | 68 (10.6) | 66.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 53 | 59 | 54 | 221
  Male | 67 | 72 | 68 | 70 | 277

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Non-Responder (NR) Participants
Description: Evaluation of the proportion of Non-Responder (NR) participants. NR correspond to the subjects who do not report any analgesic effects, with a P.I.D. (pain intensity difference) from visit 6 and visit 1 =/< 0%, (using a 0-10 NRS ). It includes the situations of average pain intensity "stable" or "worsened" at day 28 compared with baseline values.
Time Frame: 28 days
Population: Intention-to-treat
Measure: Number; unit: participants
Arm/Group | Morphine | Oxycodone | Buprenorphine | Fentanyl
Number analyzed (Participants) | 122 | 125 | 127 | 124
participants | 14 | 18 | 14 | 11

2. Secondary Outcome: Proportion of Full-responder
Description: Evaluation of the proportion of subjects who report full analgesia (full responders: FR). FR is operationally defined as a patient with a P.I.D. =/> 30% from visit 6 and visit 1 (NRS 0 to 10).
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Morphine | Oxycodone | Buprenorphine | Fentanyl
Number analyzed (Participants) | 122 | 125 | 127 | 124
participants | 89 | 90 | 95 | 88

3. Other Pre Specified Outcome: The Opioid Escalation Index
Description: The proportion of subjects with an increase of opioid daily dose > 5% compared with the basal dosage (OEI%).
Time Frame: 28 days
Measure: Number; unit: participants
Arm/Group | Morphine | Oxycodone | Buprenorphine | Fentanyl
Number analyzed (Participants) | 122 | 125 | 127 | 124
participants | 13 | 24 | 18 | 45

ADVERSE EVENTS:
Arm/Group | Morphine | Oxycodone | Buprenorphine | Fentanyl
Serious Adverse Events (participants affected / at risk) | 5/122 | 1/125 | 1/127 | 5/124
Other Adverse Events (participants affected / at risk) | 103/122 | 98/125 | 108/127 | 95/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=122) | Oxycodone (N=125) | Buprenorphine (N=127) | Fentanyl (N=124)
bowel occlusion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
exitus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
hyperalgesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
asthenia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
decline general condition (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
oral cavity bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
hyperpyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hepatic disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morphine (N=122) | Oxycodone (N=125) | Buprenorphine (N=127) | Fentanyl (N=124)
drowsiness (General disorders) | 79 (79) | 74 (74) | 81 (81) | 70 (70)
Confusion (General disorders) | 59 (59) | 55 (55) | 61 (61) | 46 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No